CLINICAL TRIAL: NCT03711994
Title: Cold Therapy for Pain Control Following Caesarean Section at Erlanger Baroness Hospital
Brief Title: Cold Therapy for Pain Control Following Caesarean Section
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to get product at this time
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-133
Record Dates: First submitted 2016-01-25; First posted 2018-10-19 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2018-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Repeat C/S Control (No Intervention): Repeat C/S done with spinal without Alkantis ice pack but with similar size dressings.
- Repeat C/S Treatment (Active Comparator): Repeat C/S done with spinal with Alkantis ice pack.
  Interventions: Other: Alkantis
- Primary C/S - Control (No Intervention): Primary C/S done with Epidural without Alkantis ice pack but with similar size dressings.
- Primary C/S Treatment (Active Comparator): Primary C/S done with Epidural with Alkantis ice pack.
  Interventions: Other: Alkantis

INTERVENTIONS:
Other: Alkantis — cold therapy pack placed on the wound post operatively
  Arms: Primary C/S Treatment; Repeat C/S Treatment

SUMMARY:
Cold Therapy has been used for a variety of procedures and has been studied in several but not recently studied for reducing postop pain following Caesarean Sections. The hypothesis is that Cold Therapy will reduce postop pain and increase patients mobility and improve care of her newborn.

DETAILED DESCRIPTION:
Cesarean Section (C/S) is one of the most commonly performed surgeries in many parts of the world. In the United States the C/S rate in 1965 was 4.5% and increased to 30.5% in 2010. While the number of C/S has increased, pain management has primarily been via epidural, spinal, local and general anesthesia and narcotic medication for the immediate postpartum period (pp). This has lead to an increase in associated cost and problems with pain management. Limited studies have been performed to evaluate cold compresses on pain relief in the immediate pp and there potential to reduce cost. Cold Therapy (CT) is most often utilized in orthopedics, sports medicine, and in general surgery. CT has been used to improve range of motion (rom) and reduce pain medication utilization. We surmise CT may be useful in decreasing narcotic utilization after C/S, as well as improve mobility and allow for improved care of the newborn. This is significant as Erlanger Baroness Hospital (EBH) is becoming Baby Friendly (BF). This is a National Initiative for Children's Healthcare Quality (NICHQ) which desires having babies rooming in with their mothers and increasing breastfeeding rates. The goal of this study is to evaluate a newer sterile delivery system for decreasing pp pain via CT. This will be done as a Randomized Controlled Trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* greater than 36 weeks gestation
* primary C/S with Epidural for labor problems or breech presentation
* Repeat C/S with spinal

Exclusion Criteria:

* less than 36.0 week gestations
* vertical skin incisions
* classical or vertical hysterotomy incisions
* failed vaginal births after C/S (VBAC)
* past history of drug or alcohol abuse
* positive drug screens unless medical prescribed drugs
* general anesthesia
* Caesarean Hysterectomy
* primary C/S with spinal anesthesia

Ages: 16 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Post Operative Pain | 48 hours after surgery
  Will Utilize Visual Analog Scales to evaluate and measure pain in the post operative period.

SECONDARY OUTCOMES:
Narcotic Utilization | 48 hours after surgrey
  Evaluate total narcotics used during time frame

CONTACTS AND LOCATIONS:
Overall Officials: William E Gist, M.D., Principal Investigator — University of Tennessee College of Medicine- Chattanooga; Kreg Jonson, M.D., Study Director — University of Tennessee College of Medicine- Chattanooga; Mandi Raper, Study Director — University of Tennessee College of Medicine- Chattanooga; Erin Tannous, MD, Study Director — University of Tennessee College of Medicine- Chattanooga; Olkayoude Akinlaja, MD, Study Chair — University of Tennessee College of Medicine- Chattanooga
Locations (1):
- Erlanger Hospital, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Placek PJ, Taffel SM. Trends in cesarean section rates for the United States, 1970--78. Public Health Rep. 1980 Nov-Dec;95(6):540-8. PMID 7433601
- [Background] Placek PJ, Taffel S, Moien M. Cesarean section delivery rates: United States, 1981. Am J Public Health. 1983 Aug;73(8):861-2. doi: 10.2105/ajph.73.8.861. PMID 6869638
- [Background] Stafford RS. Alternative strategies for controlling rising cesarean section rates. JAMA. 1990 Feb 2;263(5):683-7. PMID 2296123
- [Background] Amin-Hanjani S, Corcoran J, Chatwani A. Cold therapy in the management of postoperative cesarean section pain. Am J Obstet Gynecol. 1992 Jul;167(1):108-9. doi: 10.1016/s0002-9378(11)91638-x. PMID 1442907
- [Background] Koc M, Tez M, Yoldas O, Dizen H, Gocmen E. Cooling for the reduction of postoperative pain: prospective randomized study. Hernia. 2006 Apr;10(2):184-6. doi: 10.1007/s10029-005-0062-2. Epub 2006 Jan 24. PMID 16432641
- [Background] Kullenberg B, Ylipaa S, Soderlund K, Resch S. Postoperative cryotherapy after total knee arthroplasty: a prospective study of 86 patients. J Arthroplasty. 2006 Dec;21(8):1175-9. doi: 10.1016/j.arth.2006.02.159. PMID 17162178
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021